CLINICAL TRIAL: NCT00335855
Title: Demonstration of Safety, Effectiveness, and Ease-of-Use of an Advanced Self-Delivery System (Pharma-Pen™) for IM and SC Administration of Vaccines by Untrained Users - Phase I
Brief Title: Pharma-Pen (Formerly Innoject) Auto-injectory TIV
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-0073
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2009-04

CONDITIONS: Influenza
Keywords: Device, influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Device: Auto-injector for IM/SC vaccine administration

SUMMARY:
The purpose of this study is to evaluate the safety, effectiveness, and tolerability, of the Pharma-Pen(TM) intramuscular (IM) and subcutaneous (SC) auto-injector systems used by untrained users to self-administer Influenza vaccines as compared to standard IM injections administered by a licensed healthcare professional (e.g. a nurse). Participants will be 120 healthy men and women aged 18 - 50 years who have not received influenza vaccine for at least four years and who have no experience in giving intramuscular or subcutaneous injections. Subjects will be randomly placed in one of three treatment types. They will receive one injection of commercially available Influenza vaccine and will be evaluated over the course of six months.

DETAILED DESCRIPTION:
Pharma-Pen, Inc. (hereinafter "Pharma-Pen") and Virginia Commonwealth University ("VCU") have partnered to demonstrate the safety, effectiveness and tolerability of two versions of the Pharma-Pen(TM) auto-injector for IM injection (Treatment 1) or SC injection (Treatment 2) by untrained users compared to standard IM injection (Treatment 3) by a licensed healthcare professional (e.g. nurse). Commercially available Influenza vaccine will be used as a model to demonstrate the ease-of-use and effectiveness of the delivery system. The proposed study will compare safety and immunogenicity of three treatments in healthy volunteers: 1) Self-administered flu vaccine given IM by auto-injector in the thigh; 2) Self-administered flu vaccine given subcutaneously by auto-injector in the thigh; 3) Standard IM vaccine administered in the deltoid muscle by a licensed clinician. Primary objectives of this program are to demonstrate that the Pharma-Pen(TM) system can be safely and successfully used by untrained adults to self-inject with vaccines and to show that the resulting immunogenicity is comparable to vaccinations administered by trained medical personnel using conventional syringe/needle technology. There will be secondary information that accrues from the study. The outcomes of the IM route can be compared to the outcomes of the SC route, and the outcomes of the IM route in the deltoid muscle can be compared to the outcomes in the lateral thigh muscle. This safety/proof-of-concept study will be a randomized, single-dose, open-label, parallel, three treatment trial in 120 healthy subjects (male & female, ages 18 to 50 years) who have not received an influenza vaccine for at least four years, meet all inclusion/exclusion criteria, and sign an informed consent form. The individuals should be non-medical individuals with no experience in giving IM or SC injections. Each subject will be randomly assigned to one of three treatments. The study is divided into two successive parts (1A and 1B). Part 1A will be conducted in the first 12 subjects who will be randomized to only Treatment 1 (3 males, 3 females) and Treatment 2 (3 males, 3 females). The purpose of part 1A is to obtain initial safety information on the IM and SC auto-injectors (Pharma-Pen[TM]) in a few carefully observed subjects (10% of total) to assure that the devices are functioning as designed and do not produce significant injury to the injection site. Part 1A will be conducted under the direct supervision of the Medical Investigator (MI). The results of part 1A will be forwarded to the appointed Safety Monitoring Committee (SMC). If serious device deficiencies are detected early in part 1A, the study may be terminated prior to all 12 subjects completing this initial phase. Part 1B will be initiated only after approval of the MI and SMC, based upon the data from the 12 subjects in part 1A. Part 1B will involve the remaining 108 subjects. All injections will be performed under licensed clinician supervision.

ELIGIBILITY:
Inclusion Criteria:

1. All Subjects will be men or women between the ages of 18 and 50 years.
2. Able and willing to provide Informed Consent.
3. No previous experience of self-administered IM or SC injections.
4. In good health (no chronic diseases or medications apart from vitamins and contraceptives) as assessed by the study clinician.

Exclusion Criteria:

1. Have received influenza vaccine or had the flu in the past 4 years.
2. Have a known hypersensitivity to eggs, thimerosal or any other vaccines.
3. Subjects receiving immunosuppressive therapy within 6 weeks of enrollment.
4. Subjects who have a documented immunosuppressive syndrome.
5. Persons who have had a serious allergic reaction or other problems after exposure to influenza vaccine.
6. Persons with acute respiratory infections or other active infections or illnesses including active neurological disorders.
7. Adults with chronic metabolic diseases (including diabetes mellitus), renal dysfunction, hemoglobinopathies, or immunosuppression (including immunosuppression caused by medications or by human immunodeficiency virus [HIV]).
8. Adults who have chronic disorders of the pulmonary or cardiovascular systems, including asthma.
9. Persons with a history of Guillain-Barré syndrome (GBS).
10. Women that are pregnant or expect to become pregnant within the next 6 weeks.
11. Persons with history of thrombocytopenia or bleeding disorders.
12. Persons who have received a blood or plasma transfusion of immunoglobulin during the past 12 months.
13. Current drug abuse or alcoholism as reported by Subject.
14. History of alcohol or drug abuse in the last 5 years.
15. Have taken any immunosuppressive medications for the duration of the study.
16. Current participation in any other clinical trial or planned participation in any clinical trial in the 6 months follow-up period.
17. Subjects that state they are unable or unwilling to return to the clinic for the scheduled one month follow-up.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2006-10

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States